CLINICAL TRIAL: NCT00233935
Title: Phase Ib Randomized, Double-Blinded, Placebo-Controlled, Dose Escalation Study of Polyphenon E in Patients With Barrett's Esophagus
Brief Title: Defined Green Tea Catechin Extract in Preventing Esophageal Cancer in Patients With Barrett's Esophagus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCI-2009-00855; NCI-2009-00855 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000653460; CDR0000429486; IRB-AAAB0407; 2004-0907 (Other: Columbia University Medical Center); MDA03-1-01 (Other: DCP); N01CN35159 (NIH); P30CA013696 (NIH)
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2013-04

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — polyphenon E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm I (1 capsule) (Experimental): Patients receive 1 capsule of defined green tea catechin extract PO BID for the next 6 months.
  Interventions: Drug: defined green tea catechin extract
- Arm II (2 capsules) (Experimental): Patients receive 2 capsules of defined green tea catechin extract PO BID for the next 6 months.
  Interventions: Drug: defined green tea catechin extract
- Arm III (3 capsules) (Experimental): Patients receive 3 capsules of defined green tea catechin extract PO BID for the next 6 months.
  Interventions: Drug: defined green tea catechin extract
- Arm IV (placebo) (Placebo Comparator): Patients receive 1-3 capsules of placebo PO BID for the next 6 months.
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm IV (placebo)
Drug: defined green tea catechin extract — Given PO
  Other Names: Polyphenon E
  Arms: Arm I (1 capsule); Arm II (2 capsules); Arm III (3 capsules)

SUMMARY:
The goal of this clinical research study is to test the safety of defined green tea catechin extract at different dose levels. Researchers also want to find out what effects, good and bad, it may have on individual and their risk for esophagus cancer. Esophagus cancer is an increased risk associated with Barrett's esophagus. Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of defined green tea catechin extract may prevent esophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this study is to demonstrate the safety (i.e., determine the maximum tolerated dose (MTD)) of using Polyphenon E (Poly E) over a six-month period in the management of patients with Barrett's Esophagus (BE) with or without low-grade dysplasia (LGD).

SECONDARY OBJECTIVES:

I. To investigate the dose-related biologic effects and pharmacodynamic properties of Poly E (in order of decreasing priority):

II. Determine the efficacy of Poly E in inhibiting phosphorylation of EGFR or Her-2 or akt in esophageal mucosa.

III. Determine the pharmacodynamic profile of Poly E constituents (EGCG, EGC, EC) in esophageal tissue during and after 6 months of therapy using HPLC and GC-MS.

IV. Evaluate the efficacy of Poly E in reducing or stabilizing metaplasia and dysplasia of esophageal Barrett's mucosa using visual endoscopic measurements and histological analysis.

V. Determine the efficacy of Poly E in modulating surrogate biomarkers in esophageal mucosa - degrees of tetraploidy and aneuploidy; expression of cyclin D1, COX-2, EGFR, Her-2, akt, and Ki-67; LOH at 9p (p16) and 17p (p53); apoptotic index.

VI. Determine the efficacy of Poly E in inhibiting methylation of p16. VII. Determine the efficacy of Poly E in modulating eicosanoid levels (including PGE2) and lipoxygenase profiles in esophageal mucosa.

The esophagus is the tube used for swallowing that connects the mouth to the stomach. Barrett's esophagus is a condition in which the tissue lining of the esophagus is abnormal. It develops in some people who have heartburn, reflux disease (acid in the esophagus), or esophagitis (inflammation of the esophagus). Patients with this condition have a higher risk of developing a type of cancer of the esophagus called adenocarcinoma.

Polyphenon E (Poly E [defined green tea catechin extract]) is a low-caffeinated polyphenol mixture that is made from green tea. Poly E contains a chemical called Epigallocatechin-3 (EGCG) and other chemicals called "catechins." Research has shown that green tea, Poly E, and EGCG may be effective in preventing cancer. Poly E, as used in this study, does not contain green tea, but is made from products of green tea.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. These procedures are part of regular care for someone at increased risk of esophagus cancer. If you have had some of them recently, they may not need to be repeated. This will be up to your study doctor. You will have a complete physical exam, and your medical history will be reviewed. You will also have routine blood tests (about 2-3 tablespoons), as well as an electrocardiogram (ECG--a test to measure the electrical activity of the heart).

If you are eligible to take part in the study, and you choose to take part, you will have to complete a 1-month "wash-out period." The "wash-out period" is a period in which you must not take medications, herbs, vitamins or mineral supplements that contain tea compounds. The "wash-out" is a 30-day period before the baseline endoscopy. Because caffeine and tea may affect the results of this trial, you will be asked to not drink any tea-containing products. You will also be asked to record the amount of caffeine-containing foods and medications that you consume. You will be given a list of caffeine-containing foods and medications.

After the "wash-out" period, you will need to have a complete endoscopy and biopsy of your esophagus. This is part of regular care for someone at increased risk for esophagus cancer. This procedure will be performed in the outpatient setting. An endoscopy is an exam used by your doctor to look at your esophagus (the tube that connects your mouth and stomach) and stomach. Your doctor will place a thin scope into your mouth and carefully move the scope down the esophagus and into the stomach. During the endoscopy, you will have a standard biopsy, and a small area of abnormal tissue will be "snipped" off. The sample will be sent to the lab to look at the chemical and structural make-up of the cells of the esophageal lining. This test will be used to find out the extent of the Barrett's Esophagus.

Women who are able to have children must have a negative blood pregnancy test within 2 weeks of being assigned to a treatment group.

You will then be randomly assigned (as in a roll of the dice) by computer into one of 4 study groups. You have an equal chance of being placed in each group. Neither you nor your doctor can choose the group you will be in. Neither you, the research staff, nor your doctor will know if you are taking Poly E or placebo capsules. In this study, you will get either defined green tea catechin extract (at 1 of 3 different doses) or the placebo (a harmless drug that looks like the study drug but has no medical benefit).

If you are assigned to Group 1 ("Arm I"), you will begin taking 1 capsule of defined green tea catechin extract orally (PO) twice daily (BID) for the next 6 months.

If you are assigned to Group 2 ("Arm II"), you will begin taking 2 capsules of defined green tea catechin extract PO BID for the next 6 months.

If you are assigned to Group 3 ("Arm III"), you will begin taking 3 capsules of defined green tea catechin extract PO BID for the next 6 months.

If you are assigned to Group 4 ("Arm IV"), you will begin taking 1-3 capsules of placebo PO BID for the next 6 months. The numbers you take in this group will depend on the amount of EGCG you are assigned to receive. Each 200 mg Poly E capsule contains 200 mg of EGCG. The dosage of Poly E is based on the EGCG content. The study capsules do not contain green tea.

You will be asked to keep a study diary during your entire participation in this study. In this diary, you will record exactly when you take each dose of study drug, and how much you took each time. You will also be asked to record the amount of caffeine-containing foods and medications that you consume.

You may continue your histamine antagonist (for example, Zantac or Tagamet) or proton pump inhibitor (for example, Nexium or Prilosec) for any symptoms you may have.

Certain tests and procedures will be performed during the study, to see how the treatment is affecting your body. These tests will be done every 2 weeks for the first month, then once a month until the completion of 6 months of treatment. You will have 20-minute follow-up visits, that will including checking for any side effects and counting and writing down how much medication you have taken. You will have blood drawn (about 2-3 tablespoons) for routine tests, and you will also have urine tests (1 sample is less than 1 tablespoon).

Patients with Barrett's esophagus usually have an endoscopy every 1-3 years. For this study, it will be performed twice (at the first visit and at the 6-month visit). You will have to sign a separate consent form for each endoscopy. You cannot take aspirin, aspirin-containing substances, coumadin (warfarin), heparin, or iron supplements for 5 days before each endoscopy.

You may be taken off study if intolerable side effects occur, if the study doctor believes it is in your best interest, if you do not follow the study rules, or if the sponsor decides to stop the study for any reason.

When you have finished taking 6 months of "treatment" (either the Poly E or the placebo), you will have a follow-up endoscopy and biopsy. You will have follow-up visits scheduled for 3 months and 6 months after completing treatment. During these visits, you will be checked for side effects, blood (about 2-3 tablespoons) will be drawn for routine tests, and you will also have urine tests (1 sample is less than 1 tablespoon) performed. You will be contacted by telephone monthly after completing treatment, to check for side effects that you may be experiencing.

This is an investigational study. Poly E has been authorized for use in research only. Up to 55 participants will take part in this multicenter study. About 12 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of Barrett's metaplasia within 12 months prior to trial entry
* Note: The presence of LGD may be subject to disagreement between pathologists; this will not affect trial entry, since patients with or without LGD are eligible to participate; all cases in which there is disagreement regarding the presence of LGD will be reviewed by a third pathologist for histological classification prior to the efficacy analysis
* Cases of short-segment (less than or equal to 3 cm) Barrett's esophagus must be large enough to allow adequate sampling of tissue without completely resecting the metaplasia
* ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%)
* Leukocytes greater than or equal to 3,000/UL
* Absolute neutrophil count greater than or equal to 1,500/UL
* Platelets greater than or equal to 100,000/UL
* Total bilirubin within normal institutional limits
* AST (SGOT)/ALT (SGPT) less than or equal to institutional ULN
* Creatinine within normal institutional limits
* Alkaline phosphatase less than or equal to the institutional ULN
* Willingness to abstain from all tea consumption while on the study drug
* Willingness to record intake of caffeine-containing foods and medications while on the study
* A significant portion of caffeine intake occurs from "hidden" sources, including medications and foods
* Study subjects will be provided a list of permissible medications, beverages and foods which contain caffeine
* Participants may continue therapy with proton pump inhibitors, nonsteroidal anti-inflammatory agents, and celecoxib or rofecoxib
* Pregnancy testing to within 2 weeks prior to randomization
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* If a female participant does become pregnant while on study, she will be removed from the study
* Willingness to comply with all treatment and follow-up procedures
* Willingness to wait at least one month since last endoscopic evaluation
* Ability to understand and willingness to sign a written informed consent document
* Inclusion of women and minorities: both men and women and members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Histologically confirmed high-grade dysplasia
* Histologically confirmed diagnosis of invasive carcinoma of the esophagus
* Prior endoscopic therapy for Barrett's esophagus, including mucosal ablation, resection and esophagectomy, and photodynamic therapy
* History of esophageal strictures with moderate-to-severe dysphagia or odynophagia that may interfere with ingestion/swallowing of the study drug
* Trial participation will be determined by the study investigator after consideration of other factors including severity of dysphagia and odynophagia, necessity for treatment of strictures, and nutritional status
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Poly E
* Participants may not be receiving any other investigational agents within 30 days prior to randomization or during the study
* Use of medications, herbs, and vitamin and mineral supplements that contain tea compounds should not be taken while participating in the study and on study drug and for 30 days prior to trial entry
* If patients are consuming any of these items and would like to participate in this study, then a 30-day voluntary washout will be required
* Uncontrolled or significant co-morbid illness including, but not limited to, active or serious infection requiring intravenous antibiotics; symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia;
* Stages Ia or Ib invasive squamous cell carcinoma of the cervix treated by surgery and/or radiation therapy, stage Ia grade 1 adenocarcinoma of the endometrium treated with surgery; patients receiving active chemotherapy or radiation; or psychiatric illness/social situations that would limit compliance with study requirements
* Participants will not take aspirin, aspirin-containing substances, Coumadin (warfarin), heparin, or iron for 5 days before each endoscopy
* Active gastrointestinal bleeding; predisposing condition to gastrointestinal bleeding (including but not limited to gastritis, diverticulitis, colitis, and hemorrhoids); active malignancy diagnosed or treated within 5 years, except for squamous cell carcinoma of the skin, basal cell carcinoma of the skin, carcinoma in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Toxicity defined according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (Version 3.0) | Up to 6 months

SECONDARY OUTCOMES:
Dose-related biologic effects and pharmacodynamic properties of Poly E | Up to 6 months
  Generalized linear models will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Lightdale, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Columbia University Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - M D Anderson Cancer Center, Houston, Texas